CLINICAL TRIAL: NCT03389438
Title: A Single-center Randomized Controlled Trial of Autologous Cellular Immunotherapy in Patients With Metastatic Bladder Urothelial Carcinoma Treated With First-line Gemcitabine Plus Cisplatin
Brief Title: Autologous Cellular Immunotherapy in Patients With Metastatic Bladder Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Shortage of funds.
Sponsor: Beijing Huanxing Cancer Hospital (Other)
Collaborators: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingHCH
Record Dates: First submitted 2017-12-27; First posted 2018-01-03 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2017-12

CONDITIONS: Urinary Bladder Neoplasm
Keywords: Immunotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Experimental arm: autologous Tcm cells immunotherapy. participants who were treated with autologous Tcm cells immunotherapy.
  No intervention arm: participants who were treated with no autologous Tcm cells immunotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Participants who were treated with autologous Tcm cells immunotherapy.
  Interventions: Biological: autologous Tcm cells immunotherapy
- No intervention arm (No Intervention): Participants who were treated with no autologous Tcm cells immunotherapy.

INTERVENTIONS:
Biological: autologous Tcm cells immunotherapy — Autologous Tcm cells immunotherapy is to collect patient's own immune cells and infuse back into the patient's body after culture in vitro that can activate the anti-tumor immune response and achieve the purpose of cancer treatment.
  Arms: Experimental arm

SUMMARY:
Autologous cellular immunotherapy is to collect patient's own immune cells and infuse back into the patient's body after culture in vitro that can activate the anti-tumor immune response and achieve the purpose of cancer treatment. Central memory T (Tcm) cells are effective anti-tumor immune cells with long-term in vivo survival and self-renewal capacity. Combination of autologous Tcm cells immunotherapy with other therapies, such as surgery and chemotherapy, can effectively prolong the patient's life, prevent the recurrence and metastasis of cancers, and improve the quality of life of patients.

This study will recruit patients with pathologically and radiographically confirmed metastatic bladder urothelial carcinoma that the efficacy is evaluated as partial response (PR) or complete response (CR) after 4 cycles of the standard first-line gemcitabine plus cisplatin chemotherapy. Patients must have adequate hematologic and end-organ function, performance status and no contraindications to receive autologous Tcm cells immunotherapy. All participants will be treated with standard first-line gemcitabine plus cisplatin chemotherapy before enrolment.

This clinical trial was designed with a single-center randomized controlled trial. The study will recruit 56 patients that will be divided into treatment group and control group as 1:1 according to the randomization. Patients of treatment group will be treated with twice autologous Tcm cells immunotherapy after chemotherapy. These patients will be infused in 2-4×10^9 cells/100 ml after chemotherapy for 1 month, then cells will be infused as the same dose after another month. All patients will be followed up with hospital visits and telephone interviews to second-line treatment for disease progression. The observation period of patients is 24 months.

The objective of the study is to evaluate the clinical efficacy and safety of autologous Tcm cells immunotherapy in patients with metastatic bladder epithelial carcinoma treated with first-line gemcitabine plus cisplatin according to the progression-free survival (PFS) and overall survival (OS) of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Patients with pathologically and radiographically confirmed metastatic bladder urothelial carcinoma that the efficacy was evaluated as PR or CR after 4 cycles of the standard first-line gemcitabine plus cisplatin
3. 18-75 years old
4. CR or PR confirmed by independent radiological examination.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate hematologic and end-organ function:

   Hemoglobin ≥ 9.0g/dl, Absolute neutrophil count (ANC) > 1,500/mm3, platelets ≥ 50,000/ul Total bilirubin (TBIL) ≤ 2mg/dl, Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 the upper limit of normal (ULN) for the institution, Alkaline phosphatase (ALP) ≤ 4 the upper limit of ULN, Prothrombin time (PT) > 50% or prothrombin time-international normalized ratio (PT-INR) < 2.3, Serum creatinine (CREA) ≤ 1.5 the upper limit of ULN.
7. Qualified scanning (CT or MRI) was performed in 4 weeks before the study.

Exclusion Criteria:

1. Patients who were evaluated as stable disease (SD) or progressive disease (PD) after 4 cycles of chemotherapy.
2. Subjects with pathologically bladder urothelial carcinoma of mixed other pathological types such as squamous differentiation or sarcoma are not allowed.
3. Prior radiation therapy to the bladder
4. Significant cardiovascular disease:

   Evidence of NYHA (New York Heart Association) functional class III or IV heart disease.

   Unstable coronary artery disease (CAD) is not allowed, while Myocardial Infarction (MI) 6 months of starting study is allowed.

   Cardiac arrhythmias requiring antiarrhythmic drugs except β-blockers or digoxin are not allowed.

   Uncontrolled hypertension.
5. History of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
6. Severe infection (NCI CTCAE Version 3.0 grade > 2).
7. Subjects with epilepsy requiring steroid or antiepileptic drugs.
8. History of allotransplantation.
9. History or any evidence of hemorrhage.
10. Subjects undergoing renal dialysis.
11. Prior or undergoing cancers that primary sites are different from the cancer of this study. Exceptions to this are Cervical carcinoma in situ (CIS), Cured basal cell carcinoma and Cured cancers over 3 years before the study.
12. Ascites that is not controlled by diuretic treatment.
13. History of encephalopathy.
14. Subjects with gastrointestinal hemorrhage in 30 days before the study.
15. Subjects with history of esophageal variceal hemorrhage and it is no effective treatment to prevent the recurrence of hemorrhage.
16. Major surgery was performed in 4 weeks before the study.
17. Autologous bone marrow transplantation (ABMT) in 4 weeks before the study.
18. Concurrent treatment on another clinical trial or treatment on another clinical trial in 4 weeks before the study.
19. Pregnancy or breast-feeding.
20. There are drug abuse, medical treatment, mental illness and social disorders that would interfere with subjects' participation, or confound the results of the trial.
21. Any condition that would interfere with or endanger the safety and compliance of subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | 12 weeks
  To evaluate the clinical efficacy and safety of autologous Tcm cells immunotherapy in patients with metastatic bladder epithelial carcinoma treated with first-line gemcitabine plus cisplatin according to the progression-free survival (PFS).

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 weeks
  To evaluate the overall survival of patients after autologous Tcm cells immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, Master, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Linjun Hu, Study Chair — Beijing Huanxing Cancer Hospital
Locations (1):
- Huanxing ward, Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No